CLINICAL TRIAL: NCT03194828
Title: Leveraging Real-Time Medication Use Monitoring to Improve Adherence in Adults With Glaucoma
Brief Title: Real-time Glaucoma Medication Adherence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of sufficient recruitment
Sponsor: University of Tennessee (Other)
Collaborators: Kali Care (Unknown); Barney's Pharmacy (Unknown); Creative Care Pharmacy (Unknown); Hutton Pharmacy (Unknown); Mustang Drug (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-05074-XP
Record Dates: First submitted 2017-05-09; First posted 2017-06-21 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma
Keywords: Adherence; Mobile health; Real-time data
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring only (Active Comparator): Patients in this arm will be given a real-time medication use monitor to use in dispensing their topical glaucoma medication for 3 months
  Interventions: Behavioral: Medication monitoring only
- Monitoring and reminder (Experimental): Patients in this arm will be given a real-time medication use monitor to use in dispensing their topical glaucoma medication for 3 months and will receive an automated reminder (text or voice) when a missed dose is determined by the device's system
  Interventions: Behavioral: Medication reminder

INTERVENTIONS:
Behavioral: Medication reminder — Using the real-time data capture of the electronic device, an automated voice call or text message will be sent to active arm participants only when a missed dose is determined
  Arms: Monitoring and reminder
Behavioral: Medication monitoring only — Patients will use an electronic medication monitoring device to record their actual medication use
  Arms: Monitoring only

SUMMARY:
This study will evaluate the effectiveness of real-time data collected on patients taking topical medication to treat glaucoma. Patients will be randomized to two groups, the first of which will only use the study device to take their medication, while the second will use the study device and receive on-demand reminder messages, when necessary.

DETAILED DESCRIPTION:
Adherence to topical medications to treat glaucoma remains sub optimal; however, our understanding of this behavior remains limited due to biased measures of medication use. The Kali Drop device is a potential improvement in our ability to capture medication use in patients using dropper bottles by precisely capturing the amount dispensed in real-time. Moreover, such technology creates data that can be leveraged into driving behavior change using connected mobile technology in order to improve adherence and, ultimately, health outcomes. While evidence suggests that reminders may improve adherence to glaucoma medications, the power of doing so using real-time data has yet to be explored. This study will compare simple monitoring of patients to those who are being monitored and who receive reminder messages when the system determines one is necessary due to a missed dose.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Glaucoma diagnosis
* Prescription for a prostaglandin indicated for glaucoma
* Nonadherent (MPR<80%) in the last 3 months according to pharmacy records
* Owns and operates a mobile phone and willing to receive periodic reminder messages

Exclusion Criteria:

* Existing chronic eye condition in addition to glaucoma
* Scheduled for eye surgery in the next 90 days
* Prescription for a medication that will not fit in the device
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Adherence | From study baseline through the 3 months of the intervention
  Changes and differences in adherence to glaucoma medication between groups
Adherence follow-up | From study endpoint through the subsequent 3 months
  Changes and differences in adherence to glaucoma medication between groups after the intervention

SECONDARY OUTCOMES:
Medication self-efficacy using the 10-item Glaucoma Medication Adherence Self-Efficacy Scale | Change from baseline over the 3-month intervention
  Differences in self-reported medication-related self-efficacy between groups

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gatwood, PhD, Principal Investigator — University of Tennessee
Locations (7):
- United States (7):
  - Barney's Pharmacy, Augusta, Georgia
  - Barney's Pharmacy, Grovetown, Georgia
  - Barney's Pharmacy, Louisville, Georgia
  - Hutton Pharmacy, Blackwell, Oklahoma
  - Creative Care Pharmacy, Edmond, Oklahoma
  - Mustang Drug, Mustang, Oklahoma
  - University of Tennessee College of Pharmacy, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
No IPD